CLINICAL TRIAL: NCT01489657
Title: The Impact of Sleeve Gastrectomy Surgery in Obese Subjects on Metabolite Profiling
Brief Title: The Metabolite Profiling of Obese Subjects Before and After Sleeve Gastrectomy
Status: Withdrawn | Type: Observational
Why Stopped: The results were not significant, therfore the study ended prematurily
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, zohar landau, Head of Pediatric Endocrinology Service, Wolfson Medical Center
Other Study IDs: METPAR1
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery; Sleeve Gastrectomy; Metabolite Profiling
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective observational study is to generate further insight into the numerous metabolic adaptations associated with sleeve gastrectomy surgery in obese subjects by profiled serum metabolites before and after the surgery and integrated metabolite changes with clinical data.

DETAILED DESCRIPTION:
In the present study we examine the metabolic fluctuations of the most important amino acids and fatty acids to better understand the metabolic process in weight reduction in obese subjects that underwent sleeve gastrectomy surgery.

The availability of the tandem equipment for amino acids and fatty acids determinations for the medical system gives us an opportunity to investigate the metabolic turmoil of weight reduction seen in obese subjects after sleeve gastrectomy.

We evaluated the lipid metabolism by the measurements of the fraction of carnitine fatty acids which is the most available one because only a small blood specimen from a finger puncture is needed.

In the present study we measured the blood concentrations of monocarboxylic and dicarboxylic fatty acids bounded to carnitine, free carnitine and also free amino acids 2 weeks before the surgery while subjects eat their regular high caloric diet, one week, one month and 3 month after the procedure.

Carnitne fatty acids comprise only the tip of the iceberg of all circulating fatty acids in the blood with a roughly distribution of: triglycerides, phospholipids and cholesteryl fatty acids 4 (Lipids43-65), free fatty acids 0.6, and carnitne fatty acids 0.005 mM. Some additional amount is also circulating in lipoproteins. Even carnitine monocarboxylic fatty acids comprise around 1% of the free fatty acids and around 0.1% of all fatty compounds, the fluctuations in their concentrations probably reflect the most dynamics metabolic events because fatty acid oxidation must initiate by binding fatty acid to carnitine. The concentration of dicarboxylic carnitine fatty acids is much higher and comprises about 2% for malic carnitine and about 10% for glutaric carnitine in the total amount of free acids (http://www.hmdb.ca/). Yet, as for monocarboxylic fatty acids, a remarkable mass of dicarboxylic acids is still present as free acids.

For all carnitne acyl compounds the distribution forms have a high variability on different physiological conditions.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* Willing to undergo sleeve gastrectomy

Exclusion Criteria:

* Inability to sign the informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Bariatric Surgery Clinics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Landau, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Bariatric Surgery Clinic, Holon, Israel